CLINICAL TRIAL: NCT01529788
Title: A Double Blinded Randomized Controlled Trial to Compare the Efficacy, Time to Onset, and Duration of Two Botulinum Type A Exotoxins (Onabotulinum Toxin A and Abobotulinum Toxin A) in the Treatment of "Crow's Feet."
Brief Title: Onabotulinum Toxin Type A and Abobotulinum Toxin Type A Crow's Feet Rhytid Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Maas Clinic (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Principal Investigator, Corey S. Maas, M.D., Director, The Maas Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Medicis-Crow 4
Record Dates: First submitted 2012-02-08; First posted 2012-02-09 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Intrinsic Aging of Skin; Solar Elastosis
Keywords: abobotulinum toxin lateral orbital lines; BotoxCosmetic; Dysport; onabotulinum toxin; wrinkles; lateral orbital lines
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lateral orbital injection of Botox Cosmetic or Dysport (Active Comparator): Lateral orbital injection of either Botox Cosmetic, 10 units or Dysport, 30 units as a single dose in a randomized (right or left sides) double blind fashion in 90 consecutive subjects
  Interventions: Drug: Right lateral orbital injection of Botox Cosmetic or Dysport; Drug: Left lateral orbital injection of Botox Cosmetic or Dysport

INTERVENTIONS:
Drug: Right lateral orbital injection of Botox Cosmetic or Dysport — Right lateral orbital injection of Botox Cosmetic or Dysport (10 units and 30 units, respectively) divided among 4 injection points (0.05 mL [7.5 units] per injection point) divided among 4 injection points (0.05mL [2.5units]) on Day 0 of the study
  Other Names: Botox Cosmetic; Dysport
Drug: Left lateral orbital injection of Botox Cosmetic or Dysport — Left lateral orbital injection of Botox Cosmetic or Dysport (10 units and 30 units, respectively) divided among 4 injection points (0.05 mL [7.5 units] per injection point) divided among 4 injection points (0.05mL [2.5units]) on Day 0 of the study
  Other Names: Botox Cosmetic; Dysport

SUMMARY:
The objective of the study is to compare the time to onset of Dysport® versus Botox® in the treatment of lateral orbital rhytids ("crow's feet"). Thirty subjects were enrolled in the study; specifically 30 male or female patients 18 years or older with moderate to severe lateral orbital rhytids at maximum contracture. Each patient were randomized to be treated with Dysport® on one side and Botox® on the other side. Both the injector and patient were blinded to the injected toxin.

The efficacy endpoints were determined by investigator and subject live assessment of "crow's feet" at rest and maximum contraction at each visit (every other day for 6 days post-injection, every month for 9 months following) using a validated 5 point photographic scale(no wrinkles [0], very fine wrinkles [1], fine wrinkles [2], moderate wrinkles [3] or severe wrinkles [4]) used in previous studies. A written description of each photograph was included to help standardize the application of the Photographic Scale.

DETAILED DESCRIPTION:
INTRODUCTION:

Dysport® (Medicis, Scottsdale, AZ) is the formulation (previously known as 52120 and Reloxin®) of Clostridium botulinum type A (BoNT-A) toxin-hemagglutinin complex to be used in the United States (US) cosmetic clinical program. It is identical to the Ipsen product marketed outside the United States and under clinical studies in the United States for cosmetic and non-cosmetic use. Dysport® injections are used to relax the musculature of the upper face, reducing the appearance of dynamic rhytids. Previously FDA-approved Botulinum type A toxins have been utilized in the upper face to treat glabellar rhytids for nearly two decades. Botox® Cosmetic (Allergan, Irvine, CA), is the first FDA-approved Botulinum toxin type A to be approved in the United States for the treatment of glabellar rhytids. Its efficacy and safety have been proven in multiple studies. However, no comparison to onset of action exists amongst the different BoNT-A products. This study seeks to compare the onset of action between two BoNT-A products, Dysport® and Botox® Cosmetic.

BACKGROUND:

Relaxation of facial musculature is routinely accomplished for cosmetic use by the use of Clostridium botulinum type A. Clostridium botulinum type A toxin reduces the recruitment of specific muscle groups. Many studies have been published in peer-reviewed medical journals regarding the cosmetic use of this biologic.2-11 Clostridium botulinum in the form of Botox® Cosmetic is FDA-approved for cosmetic use in the treatment of rhytids in the glabellar region. Dysport®, the brand name of the Ipsen product marketed outside the United States and under clinical studies in the United States for cosmetic and non-cosmetic use, and the current name now used under FDA-approval.

Many studies have demonstrated the effect of botulinum toxin on facial rhytids produced by underlying coordinated muscle groups. Those of the glabellar area, upper forehead, lower forehead, periocular and perinasal area are particularly well-documented. Previous reports of Dysport® and Botox® Cosmetic medications show effective relaxation of glabellar rhytids after injection.12-17

The most common adverse event (AE) seen following the use of Dysport® or Botox® Cosmetic for the treatment of blepharospasm is ptosis. Some patients have reported diplopia or symptoms resulting from the spread of effect to mid-facial muscles. Other AEs reported were injection site reaction, skin rashes, influenza-like symptoms, dry eyes, tearing, bruising, and eyelid swelling. Reversible ophthalmoplegia has been reported after excessive dosing.

Multiple Phase II and III clinical studies have been conducted in North America to determine the optimal dosing of Dysport® for cosmetic use in the glabellar area, and 50 units of Dysport® is generally recognized as the optimal dosage for treatment of the glabellar region. Dysport® to Botox® Cosmetic dosing is generally a 2.5:1 or 3:1 unit for unit conversion. For the crows feet area, 10 units of Botox® Cosmetic at 4 injection points is used in a similar fashion, producing comparable results to 25 units of Dysport® at the same four injection points. What is not clear is whether one of these BoNT-A provide a quicker onset to action. This study intends to compare onset of action of both of these BoNT-A by daily live assessments of patients in the week following injection of either Dysport® or Botox® Cosmetic.

INVESTIGATIONAL AGENTS:

Dysport® is the formulation (previously known as 52120 and Reloxin®) of Clostridium botulinum type A toxin-hemagglutinin complex to be used in the United States (US) cosmetic clinical program. Reloxin® is identical to Dysport, the brand name of the Ipsen product marketed outside the United States and under clinical studies in the United States for cosmetic and non-cosmetic use.

Dysport® will be supplied as a white, lyophilized powder containing 500 units of Clostridium botulinum type A toxin-hemagglutinin complex, 125 μg human serum albumin, and 2.5 mg of lactose. Study medication will be reconstituted at the investigational center with sterile physiological saline for injection without preservative.

Botox® Cosmetic is supplied as a 100 unit vial of Clostridium botulinum type A exotoxin, sterilely prepared and vacuum-dried without preservatives. The vial also contains 0.5mg of albumin (human) and 0.9 mg of sodium chloride.

DOSE RATIONAL AND RISKS/BENEFITS:

Eligible patients will receive Dysport® (25 units) divided among 4 injection points (0.05 mL [6.25 units] per injection point) in the lateral orbital rhytid on one side and Botox® Cosmetic (10 units) divided among 4 injection points (0.05mL [2.5 units]) in the lateral orbital rhytid region on the contralateral side on Day 0 of the study.

For Study Purposes:

• For study purposes, only one injection session will be performed at Day 0 of the study. Subsequent follow-up visits will only monitor the effects of the single injection session at time 0.

Packaging, Labeling, and Storage Active drug (Dysport®) vials, bearing a unique lot number, will be sent from Ipsen Biopharm Ltd. or Medicis Pharmaceutical Corporation. Each vial will be labeled with a batch/lot number and unique sequential pack number. Beaufour Ipsen Industrie SAS will perform packaging and labeling of study medication vials in compliance with all regulatory requirements.

Unused vials will be returned to Almedical or Medicis for final accounting and destruction.

Active drug (Botox® Cosmetic) vials, bearing a unique lot number, will be sent from Allergan Inc, Irvine CA. Each vial will be labeled with a batch/lot number and unique sequential pack number.

Study medications must be maintained during transit and storage within a temperature range of 2o to 8oC. Until dispensed to the patients, study medication will be stored refrigerated in a secure location, separated from normal hospital/practice stocks, and accessible only to authorized personnel.

Reconstitution Techniques Following the dilution instructions below, the investigator (or trained designee) can prepare the individual patient's study dose for injection.

Each patient's dose will be prepared as an isovolumic (0.2 mL of normal saline) of BotoxCosmetic or Dysport injection for administration by the investigator.

Drug accountability The investigator will be supplied with a sufficient amount of study medications and confirm receipt of all batches of study medication in writing.

The investigator will administer study medication only to patients included in this study and following the procedures set out in this study protocol. Each dispensing will be documented in the CRFs and the study medication dispensing log.

Concomitant Medications and Treatments Any medication the patient takes other than the study medication specified in the protocol is considered a concomitant medication. This applies to prescription and over-the-counter (OTC) drugs, and to herbal supplements, whether taken systemically or applied topically. In addition, any treatment the patient receives other than the study medication is considered a concomitant treatment. This applies to cosmetic treatments of the face and neck area. All concomitant medications and concomitant treatments must be reco0rded in the CRFs.

Prohibited medication classes and treatments are described under "Exclusion Criteria". In the event that a prohibited treatment (e.g. microdermabrasion, Intense Pulse Light, light-emitting diodes, or radio-frequency) is received, it must be documented on the CRFs.

STUDY OBJECTIVES:

Primary Objective:

To compare the time to onset of action, efficacy and duration of Dysport® versus Botox® Cosmetic in the treatment of lateral orbital rhytids.

Secondary Objective:

To determine the safety and presence of any adverse effects of Dysport® (25 units) versus Botox® Cosmetic (10 units) in the treatment of lateral orbital rhytids.

STUDY PROCEDURES:

Visit 1 (Initial Visit and treatment day 0) This visit will serve as both screening and baseline. During this visit, the subject will receive the ICF and be consented in accordance to this site's consenting SOP. After consenting, inclusion and exclusion criteria will be obtained. If the subject meets these, then demographic data will be taken as well as clinical history and concomitant medications. The P.I. will then decide if the subject is to be included or excluded using the inclusion exclusion criteria, clinical history, visual examination of the head and neck, and concomitant medications. If the patient has the need for a pregnancy test, a urine pregnancy test will be performed in office. Assignment of patient # will occur as will randomization to receive Dysport® and Botox® Cosmetic in each lateral orbital area. The subject will then be photographed using the Canfield Digital photography system. The subject will provide a self-assessment of lateral orbital rhytids at rest using a static 5-point categorical scale. The investigator will assess in person lateral orbital rhytids at maximal contraction and at rest and lateral orbital rhytids according to a static 5-point Photographic scale validated in prior studies. Following the rating scales, the patient will be administered Dysport® to the lateral orbital area on one side and Botox® Cosmetic to the contralateral lateral orbital area (as described in Appendix 1 and Section 5.4). The patient is to remain for 30 minutes after injection to monitor for any AEs. A follow-up appointment at day 1 will be scheduled.

Visit 2 (Day 2) This visit will be a follow up at day 2. The subject will complete a form on adverse events following Dysport® or Botox® Cosmetic injection as well as the Concomitant medications/Procedures/Treatments form. The subject will then be photographed using the Canfield Digital photography system. The subject will provide a self-assessment of to the lateral orbital rhytids at rest using a static 5-point categorical scale. The investigator will assess in person lateral orbital rhytids at maximal contraction and at rest and rate lateral orbital rhytids according to a static 5-point Photographic scale. A follow-up appointment at day 4 will be scheduled.

Visit 3 (Day 4) This visit will be a follow up at day 4. The subject will complete a form on adverse events following Dysport® or Botox® Cosmetic injection as well as the Concomitant medications/Procedures/Treatments form. The subject will then be photographed using the Canfield Digital photography system. The subject will provide a self-assessment of lateral orbital rhytids at rest using a static 5-point categorical scale. The investigator will assess in person lateral orbital rhytids at maximal contraction and at rest and rate lateral orbital rhytids according to a static 5-point Photographic scale. A follow-up appointment at day 6 will be scheduled.

Visit 4 (Day 6) This visit will be a follow up at day 6. The subject will complete a form on adverse events following Dysport® or Botox® Cosmetic injection as well as the Concomitant medications/Procedures/Treatments form. The subject will then be photographed using the Canfield Digital photography system. The subject will provide a self-assessment of lateral orbital rhytids at rest using a static 5-point categorical scale. The investigator will assess in person lateral orbital rhytids at maximal contraction and at rest and rate lateral orbital rhytids according to a static 5-point Photographic scale. A follow-up appointment at day 30 will be scheduled.

Visit (Day 30),Visit 6 (Day 90),Visit 7 (Day 120),Visit 8 (Day 150),Visit 9 (Day 180), Visit 10 (Day 210), Visit 11 (Day 240), and Visit 12 (Day 270):

This visit will be a follow up at days 30, 60, 90, 120, 150, 180, 210, and 240. The subject will complete a form on adverse events following Dysport® or Botox® Cosmetic injection as well as the Concomitant medications/Procedures/Treatments form. The subject will then be photographed using the Canfield Digital photography system. The subject will provide a self-assessment of lateral orbital rhytids at rest using a static 5-point categorical scale. The investigator will assess in person lateral orbital rhytids at maximal contraction and at rest and rate lateral orbital rhytids according to a static 5-point Photographic scale. A follow-up appointment at day 90 will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients who meet all of the following criteria are eligible for this study:

* Eighteen years of age or older.
* Moderate to severe lateral orbital rhytids at maximum smile (score of [2] or [3] by physician assessment)
* Negative pregnancy test for females of childbearing potential.
* Time and ability to complete the study and comply with instructions.
* Understanding of the study and contents of the informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study:

* Previous treatment to the glabellar area, forehead or lateral orbital rhytids with Dysport® or Botox® Cosmetic or other botulinum toxin within 180 days of entry into the study. Botulinum toxin treatment of areas other than the lateral orbital rhytids at any time during the study.
* Patients with an ongoing treatment-related AE from any Dysport® or Botox® Cosmetic or botulinum toxin study.
* Inability to substantially lessen lateral orbital lines by physically spreading them apart.
* Permanent or semi-permanent dermal fillers in the lateral orbital rhytids at any time.
* Ablative skin resurfacing on the lateral orbital rhytids at any time preceding the study or planning to during the current study.
* Upper eyelid blepharoplasty or brow lift at any time preceding the study or planning to during the current study.
* Non-ablative treatments in the lateral orbital region for skin dyschromias (e.g. Intense Pulsed Light, light-emitting diodes) at any time during the current study.
* Non-ablative dermal treatment in the lateral orbital area for skin tightening (e.g. radiofrequency treatments at any time preceding the current study or planned to have this done during the current study.
* Retinoid, microdermabrasion, or prescription-level glycolic acid treatments to the lateral orbital area within 2 weeks prior to study participation or during the current study.
* Concurrent therapy that, in the investigator's opinion, would interfere with evaluation of the efficacy or safety of the medication.
* Active infection of the lateral orbital area (e.g. acute acne lesions or ulcers).
* Pregnant women, nursing mothers, or women who are planning pregnancy during the study, or think they may be pregnant at the start of the study. Throughout the course of the study, women of childbearing potential must use reliable forms of contraception (e.g. abstinence, oral contraceptives for more than 12 consecutive weeks prior to enrollment, or spermicide and condoms).
* Current history of chronic drug or alcohol abuse.
* Enrollment in any active study involving the use of investigational devices or drugs.
* Current facial palsy.
* Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
* Neuromuscular junctional disorders (myasthenia gravis).
* Known allergy or hypersensitivity to any botulinum toxin or any component of Dysport® or Botox® Cosmetic.
* Clinically diagnosed anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that, in the opinion of the investigator, might interfere with the patient's participation in the study.
* Concurrent use of medications that affect neuromuscular transmission, such as curare-like depolarizing agents, lincosamides, polymyxins, anticholinesterases affecting the striated muscle, and aminoglycoside antibiotics.
* Presence of any condition( e.g. neuromuscular disorder or other disorder that could interfere with neuromuscular function) or circumstance that, in the judgment of the investigator, might increase the risk to the patient or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To compare the time to onset of action, efficacy and duration of Dysport® versus Botox® Cosmetic in the treatment of lateral orbital rhytids. | 9 months
  Subject and investigator assessed grading as well as subject preference

SECONDARY OUTCOMES:
To determine the safety and presence of any adverse effects of Dysport® (25 units) versus Botox® Cosmetic (10 units) in the treatment of lateral orbital rhytids. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Corey S Maas, MD, Principal Investigator — The Maas Clinic
Locations (1):
- The Maas Clinic, San Francisco, California, United States

REFERENCES:
- [Background] Elson ML. Evaluation and treatment of the aging face. In: Evaluation and Treatment of the Aging Face. Elson MD, ed. Springer-Verlag, New York, 1995, 1-9.
- [Background] Lowe NJ. Botulinum toxin type A for facial rejuvenation. United States and United Kingdom perspectives. Dermatol Surg. 1998 Nov;24(11):1216-8. doi: 10.1111/j.1524-4725.1998.tb04100.x. PMID 9834741
- [Background] Guerrissi J, Sarkissian P. Local injection into mimetic muscles of botulinum toxin A for the treatment of facial lines. Ann Plast Surg. 1997 Nov;39(5):447-53. doi: 10.1097/00000637-199711000-00002. PMID 9374139
- [Background] Foster JA, Barnhorst D, Papay F, Oh PM, Wulc AE. The use of botulinum A toxin to ameliorate facial kinetic frown lines. Ophthalmology. 1996 Apr;103(4):618-22. doi: 10.1016/s0161-6420(96)30644-1. PMID 8618761
- [Background] Guyuron B, Huddleston SW. Aesthetic indications for botulinum toxin injection. Plast Reconstr Surg. 1994 Apr;93(5):913-8. doi: 10.1097/00006534-199404001-00003. PMID 8134483
- [Background] Blitzer A, Brin MF, Keen MS, Aviv JE. Botulinum toxin for the treatment of hyperfunctional lines of the face. Arch Otolaryngol Head Neck Surg. 1993 Sep;119(9):1018-22. doi: 10.1001/archotol.1993.01880210108015. PMID 8357583
- [Background] Carruthers JD, Carruthers JA. Treatment of glabellar frown lines with C. botulinum-A exotoxin. J Dermatol Surg Oncol. 1992 Jan;18(1):17-21. doi: 10.1111/j.1524-4725.1992.tb03295.x. PMID 1740562
- [Background] Fagien S. Botox for the treatment of dynamic and hyperkinetic facial lines and furrows: adjunctive use in facial aesthetic surgery. Plast Reconstr Surg. 1999 Feb;103(2):701-13. doi: 10.1097/00006534-199902000-00055. PMID 9950563
- [Background] Ramirez AL, Reeck J, Maas CS. Botulinum toxin type B (MyoBloc) in the management of hyperkinetic facial lines. Otolaryngol Head Neck Surg. 2002 May;126(5):459-67. doi: 10.1067/mhn.2002.124706. PMID 12075218
- [Background] Kim EJ, Ramirez AL, Reeck JB, Maas CS. The role of botulinum toxin type B (Myobloc) in the treatment of hyperkinetic facial lines. Plast Reconstr Surg. 2003 Oct;112(5 Suppl):88S-93S; discussion 94S-97S. doi: 10.1097/01.PRS.0000082197.88799.84. PMID 14504489
- [Background] Carruthers JA, Lowe NJ, Menter MA, Gibson J, Nordquist M, Mordaunt J, Walker P, Eadie N; BOTOX Glabellar Lines I Study Group. A multicenter, double-blind, randomized, placebo-controlled study of the efficacy and safety of botulinum toxin type A in the treatment of glabellar lines. J Am Acad Dermatol. 2002 Jun;46(6):840-9. doi: 10.1067/mjd.2002.121356. PMID 12063480
- [Background] Ascher B, Klap P, Marion MH, Chanteloub F. [Botulinum toxin in the treatment of frontoglabellar and periorbital wrinkles. An initial study]. Ann Chir Plast Esthet. 1995 Feb;40(1):67-76. French. PMID 7668808
- [Background] Ascher B. Facial rejuvenation by non-endoscopic lifting and botulinum toxin injection. Les Cahiers D'Ophthalmologie 2000;45:25-31.
- [Background] Olver JM. Botulinum toxin A treatment of overactive corrugator supercilii in thyroid eye disease. Br J Ophthalmol. 1998 May;82(5):528-33. doi: 10.1136/bjo.82.5.528. PMID 9713061
- [Background] Erian A, Ionescu NE. Combination treatment of glabellar rhytids. Int J Cosmetic Surg 1999;7(1):14-17.
- [Background] Feller G, Bayerl C, Jung E, Rzany B. Treatment of dynamic facial wrinkles with botulinum toxin type A (Dysport®)-a pilot study. Akt Deramtol 2000;26:65-9.
- [Background] Le Louarn C. [Botulinum toxin and facial wrinkles: a new injection procedure]. Ann Chir Plast Esthet. 1998 Oct;43(5):526-33. French. PMID 9882892
- [Background] Altman DG. How large a sample? Statistics in Practice. London, UK: British Medical Association 1982.
- [Background] McLarty JW, Levine RJ. How many subjects are required for a study? IRB. 1987 Sep-Oct;9(5):1-3. No abstract available. PMID 11649896